CLINICAL TRIAL: NCT00530205
Title: An Observation of the Change in Percent Lean Body Mass of Stage III Non-Small Cell Lung Cancer Undergoing Radiation Treatment
Brief Title: Effects of Radiation Therapy on the Body in Patients With Stage III Non-Small Cell Lung Cancer
Status: Withdrawn | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Jessica Stauffer, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Other Study IDs: CASE5506; P30CA043703 (NIH); CASE5506 (Other: Case Comprehensive Cancer Center); CASE-5506-CC217
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Lung Cancer; Malnutrition; Weight Changes
Keywords: weight changes; malnutrition; stage III non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Malnutrition; Body Weight Changes; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: physiologic testing
Other: questionnaire administration
Procedure: management of therapy complications
Radiation: radiation therapy

SUMMARY:
RATIONALE: Learning about the effects of radiation therapy on the body's muscles, organs, and bones in patients with stage III non-small cell lung cancer may help doctors plan the best treatment.

PURPOSE: This clinical trial is studying the effects of radiation therapy on the body in patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine energy and protein consumption on an average radiotherapy treatment day using the multiple pass method 24-hour analysis of food recall at baseline and treatment end.
* To compare energy and protein by mouth intake from baseline to treatment end.
* To measure and compare diet quality from baseline to radiotherapy treatment end by Healthy Eating Index (HEI) score.
* To determine lean body mass versus fat mass using a bioelectrical impedance analysis machine.
* To compare body fat to lean body mass percentage at baseline with that at radiotherapy treatment end.
* To correlate energy and protein consumption with lean body mass at baseline and treatment end.
* To determine the change in appetite throughout radiotherapy by comparing data obtained by interview at baseline and radiotherapy treatment end.
* To determine the change in performance level (Karnofsky percentage) associated with the radiotherapy through a series of questions asked at baseline and treatment end.

OUTLINE: Patients receive radiotherapy as planned for 7 weeks. Patients undergo an interview on treatment day 1 (before initiation of radiotherapy) and treatment day 35 (after completion of radiotherapy) regarding recent food consumption history and appetite. Patients' standing weight and height are measured on these days and their body composition, measured with a bioelectrical impedance analysis (BIA) device, are also taken. Patients' Karnofsky performance score are obtained from their medical record.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with stage III non-small cell lung cancer (NSCLC)
* Plan to begin radiotherapy for NSCLC

  * Radiotherapy is the only planned therapy for this cancer
* No brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Must be able to stand without assistance

Exclusion criteria:

* Unable to comply with study requirements
* Native language other than American English
* Pacemaker or implanted defibrillator

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Receiving chemotherapy in combination with radiotherapy
* Concurrent megace or steroids

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care center
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-02

PRIMARY OUTCOMES:
Energy and protein consumption measured on an average radiotherapy treatment day by multiple pass method 24-hour analysis for food recall at baseline and treatment end
Comparison of energy and protein by mouth intake from baseline to treatment end
Comparison of diet quality as measured by Healthy Eating Index (HEI) score from baseline to treatment end
Lean body mass versus fat mass using a bioelectrical impedance analysis machine
Comparison of body fat to lean body mass percentage at baseline and at treatment end
Correlation of energy and protein consumption with lean body mass at baseline and treatment end
Change in appetite throughout radiotherapy determined by interview at baseline and end of treatment
Change in performance level (Karnofsky percentage) associated with the radiotherapy procedure determined by questions asked at baseline and end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Stauffer, BS, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=case5506